CLINICAL TRIAL: NCT05189717
Title: A Single-arm, Open-label and Multi-center Phase I Study on Safety, Tolerance and Pharmacokinetics of HRS-8080 Tablets Monotherapy and Combined With Other Anti-cancer Therapy in Patients With Metastatic or Local Advanced Breast Cancer
Brief Title: A Trial of HRS-8080 Tablets in Metastatic or Local Advanced Breast Cancer of Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8080-I-101
Record Dates: First submitted 2021-12-16; First posted 2022-01-12 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Metastatic or Local Advanced Breast Cancer of Patients
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: HRS-8080 tablets monotherapy and combined with other anti-cancer therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group (Experimental): Firstly Dose Escalation and Dose Expansion of HRS-8080 monotherapy should be conducted. After RP2D and MTD of the HRS-8080 monotherapy were confirmed, Dose Escalation and Dose Extension of HRS-8080 in combination with other anti-cancer treatment would be completed, including SHR 6390, or Abemaciclib, or Everolimus.
  Interventions: Drug: HRS-8080 tablets、SHR 6390 tablets、Abemaciclib、Everolimus

INTERVENTIONS:
Drug: HRS-8080 tablets、SHR 6390 tablets、Abemaciclib、Everolimus — During HRS-8080 monotherapy period, the dose of HRS-8080 would be increasing. In the combination therapy period, HRS-8080 will be administered at flat dose of RP2D-1 and RP2D.

SUMMARY:
The study is being conducted to evaluate the tolerance, and safety of HRS-8080 tablets monotherapy and combined with other anti-cancer therapy for metastatic or local advanced breast cancer in adults. To explore the reasonable dosage of HRS-8080 tablets for metastatic or local advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status score: 0-1;
2. Histopathologically documented local advanced or metastatic breast cancer ;
3. Female of not childbearing potential must the related requirement;
4. During or after the last systematic therapy before enrolment, disease progression occurred with clinical or radiographical documentation;
5. Adequate organ functions as defined;
6. Ability to understand and voluntarily agrees to participate by giving written informed consent for the study.

Exclusion Criteria:

1. For the case of symptomatic visceral metastasis, the investigators judged that it was not suitable to use relevant treatment;
2. patients with active brain metastasis (without medical control or with clinical symptoms), cancerous meningitis, spinal cord compression, or patients with a history of primary tumors of the central nervous system ;
3. History of clinically significant cardiovascular or cerebrovascular diseases;
4. The subject has one of many factors affecting oral drugs;
5. Active infection or fever with unknown cause > 38.5 °C;
6. Active autoimmune diseases, History of immunodeficiency, including positive HIV serum test result and other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
7. Known history of allergy to study drug ingredients.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | up to 28 days
  The Maximum tolerated dose of HRS-8080 monotherapy or in combination with SHR-6390 / Abemaciclib / Everolimus
Recommended phase II dose | up to 28 days
  The Recommended phase II dose of HRS-8080 monotherapy or in combination with SHR-6390 / Abemaciclib / Everolimus
Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) | up to 30 days after the last dose
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) graded by Common Terminology Criteria for Adverse Events (CTCAE) v5.0

SECONDARY OUTCOMES:
Cmax | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fifth treatment period
  PK parameters of multiple doses of HRS-8080 monotherapy. HRS-8080 in combination therapy, SHR-6390, Abemaciclib and Everolimus.
Tmax | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fifth treatment period
  PK parameters of multiple doses of HRS-8080 monotherapy. HRS-8080 in combination therapy, SHR-6390, Abemaciclib and Everolimus. etc.
AUC0-t | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fifth treatment period
  PK parameters of multiple doses of HRS-8080 monotherapy. HRS-8080 in combination therapy, SHR-6390, Abemaciclib and Everolimus.
Cmax,ss | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fifth treatment period
  PK parameters of multiple doses of HRS-8080 monotherapy. HRS-8080 in combination therapy, SHR-6390, Abemaciclib and Everolimus.
Tmax,ss | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fifth treatment period
  PK parameters of multiple doses of HRS-8080 monotherapy. HRS-8080 in combination therapy, SHR-6390, Abemaciclib and Everolimus.
Cmin,ss | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fifth treatment period
  PK parameters of multiple doses of HRS-8080 monotherapy. HRS-8080 in combination therapy, SHR-6390, Abemaciclib and Everolimus.
AUCss | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fifth treatment period
  PK parameters of multiple doses of HRS-8080 monotherapy. HRS-8080 in combination therapy, SHR-6390, Abemaciclib and Everolimus.
Rac | 0.5 hour before first dose of first treatment period to the 0.5 hour before first dose of fifth treatment period
  PK parameters of multiple doses of HRS-8080 monotherapy. HRS-8080 in combination therapy, SHR-6390, Abemaciclib and Everolimus.
ORR | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 8 months
  Objective Response Rate, Preliminary Efficacy endpoints of HRS-8080 monotherapy or in combination with SHR-6390, Abemaciclib or Everolimus in treatment of patients with metastatic or local advanced breast cancer
BOR | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 8 months
  Best Overall Response, Preliminary Efficacy endpoints of HRS-8080 monotherapy or in combination with SHR-6390, Abemaciclib or Everolimus in treatment of patients with metastatic or local advanced breast cancer
DoR | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 8 months
  Duration of response, Preliminary Efficacy endpoints of HRS-8080 monotherapy or in combination with SHR-6390, Abemaciclib or Everolimus in treatment of patients with metastatic or local advanced breast cancer
DCR | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 8 months
  Disease control rate, Preliminary Efficacy endpoints of HRS-8080 monotherapy or in combination with SHR-6390, Abemaciclib or Everolimus in treatment of patients with metastatic or local advanced breast cancer
PFS | from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 8 months
  Progression-free survival, Preliminary Efficacy endpoints of HRS-8080 monotherapy or in combination with SHR-6390, Abemaciclib or Everolimus in treatment of patients with metastatic or local advanced breast cancer

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Fifth Medical Center of People's Liberation Army of China General Hospital, Beijing, Beijing Municipality
  - Jilin Cancer Hospital, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: Undecided